CLINICAL TRIAL: NCT04879017
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation and Expansion Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Orally Administered FHD-286 in Subjects With Metastatic Uveal Melanoma
Brief Title: FHD-286 in Subjects With Metastatic Uveal Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated the study for business reasons.
Sponsor: Foghorn Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FHD-286-C-001
Record Dates: First submitted 2021-04-28; First posted 2021-05-10 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Uveal Melanoma
Keywords: UM; metastatic uveal melanoma; advanced uveal melanoma; phase 1; FHD-286; Foghorn
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Intervention Model Description: Open label single arm dose escalation and two-arm expansion study in patients with metastatic UM
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FHD-286 dose escalation and expansion (Experimental): Up to approximately 125 patients will be enrolled in dose escalation and expansion
  Interventions: Drug: FHD-286

INTERVENTIONS:
Drug: FHD-286 — FHD-286 as a single agent

SUMMARY:
This Phase 1, multicenter, open-label, dose escalation and expansion study is designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of FHD-286 oral monotherapy in subjects with metastatic Uveal Melanoma (UM).

DETAILED DESCRIPTION:
This study is an ascending multiple dose clinical trial with expansion arms. It is primarily intended to evaluate the safety and tolerability of FHD-286 when administered orally to subjects with metastatic UM. The Dose Escalation Phase will allow for the determination of the recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) in subjects with metastatic UM. This study will also evaluate the PK/PD profiles of multiple dose administration of FHD-286.

The Dose Expansion Phase will allow a more robust evaluation of the safety profile of FHD-286, including less frequent toxicities and an assessment of antitumor activity. The data from this study in subjects with metastatic UM, including safety, tolerability, PK/PD findings, and antitumor activity, will form the basis for subsequent clinical development of FHD-286.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects ≥ 18 years of age
* Subject must have a diagnosis of metastatic histologically or cytologically confirmed UM. If histologic or cytologic confirmation of the primary tumor is not available, clinical confirmation of a diagnosis of metastatic UM, as per standard practice for UM, by the treating investigator can be obtained, and fall into any of the following categories:

  1. Newly diagnosed subject who has not yet received liver-directed or systemic treatment
  2. Subjects ineligible for any available therapy likely to convey clinical benefit
  3. Subjects who have disease progression after treatment with available therapies and/or who is intolerant to those treatments.
* Subject must have measurable disease by RECIST v1.1, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) as ≥ 10 mm with calipers and/or CT scan. Measurable lesions cannot have undergone any local treatment (including liver-directed radio- or immune-therapies) or radiation, unless there has been interim progression of that lesion, nor can any local treatment or radiation involving measurable lesions be anticipated.

Note: A malignant lymph node must be ≥ 15 mm on the short axis when assessed by CT scan to be considered pathologically enlarged and measurable.

* Willingness to provide newly obtained tumor tissue at baseline and on treatment unless contraindicated by medical risk in the opinion of the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 2. a.) Arm 2 (Dose Expansion Phase): Subjects enrolling in Arm 2 must have an ECOG PS of ≤ 3.

Key Exclusion Criteria:

* Subjects who have other malignancy which may interfere with the diagnosis and/or treatment of metastatic UM.
* Subject has thrombocytopenia (platelets < 50 × 109/L) or another major bleeding disorder/diathesis.

Note: Subjects with platelets < 50 × 109/L may be permitted to enroll only in Arm 2 of the Dose Expansion Phase at the discretion of the Investigator and the Sponsor.

* Subject has active brain metastases and/or leptomeningeal disease. Subjects with known CNS metastases are only permitted under the following conditions; exceptions may be made on a case-by-case basis with the approval of the Sponsor: Brain metastases must have been stable for approximately 2 months since completion of most recent CNS-directed intervention. Subject may be on corticosteroids so long as the dose is stable for approximately 14 days or decreasing at the time of study entry. Anti-epileptic therapy is allowed so long as medications are not otherwise excluded and seizures have been controlled for approximately 4 weeks since last anti-epileptic medication adjustment.

  1. Dose Escalation Phase: Subjects with known CNS metastases that meet the above conditions are permitted to enroll in dose escalation.
  2. Arm 1 (Dose Expansion Phase): Subjects with known or suspected CNS metastases are excluded from Arm 1.
  3. Arm 2 (Dose Expansion Phase): Subjects with CNS metastases that meet the above conditions are permitted to enroll in Arm 2.
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections; subjects with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Subject has known positive HIV antibody results or acquired immunodeficiency syndrome (AIDS)-related illness; subjects with CD4+ T-cell counts greater than or equal to 350 cells/µL will be permitted, as will subjects who have not had an AIDS-related illness within the past 12 months
* Subjects with an active infection cannot be enrolled until any required antibiotic and/or antifungal therapy has been completed and/or infection is determined to be controlled
* Subjects who have an uncontrolled intercurrent illness.
* Known and possible risk for QT prolongation.
* Subject is on medications that are strong CYP3A inhibitors, are strong CYP3A inducers, or are sensitive CYP3A substrates with narrow TIs
* Subject is on medications with narrow TIs that are sensitive P-gp or BCRP substrates and are administered orally such as digoxin
* Subjects who require clinically significant or increasing doses of systemic steroid therapy or any other systemic immunosuppressive medication. The use of a stable dose of systemic steroids and/or immunosuppressive medication is permitted with Sponsor approval. Local or targeted steroid and immunosuppressive therapies (e.g. inhaled or topical steroids) are acceptable. Appropriate steroid replacement to manage endocrine toxicities resulting from prior systemic anticancer therapy is permitted. See exclusion criterion 3 for exceptions regarding steroid therapy for subjects with CNS metastases. See exclusion criterion 13 for exclusions regarding medications that are strong CYP3A inhibitors, strong CYP3A inducers, or sensitive CYP3A substrates with narrow TIs.
* Subjects have undergone any prior treatment with a BRG1/BRM inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 31 months
  Dose escalation and expansion
Incidence of adverse events (AEs), serious adverse events (SAEs) including changes in safety laboratory parameters and AEs leading to discontinuation | Up to 31 months
  Dose escalation and expansion
Incidence of dose limiting toxicities (DLTs) during cycle 1 (28 days) | Cycle 1 (cycle length = 28 days)
  Dose escalation

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 30 months
  ORR is defined as the percentage of subjects with evidence of a complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.
Duration of Response (DOR) | Up to 30 months
  DOR is defined as the time from first documented evidence of CR or PR until the earliest date of documented radiological progression per RECIST 1.1. or death due to any cause among subjects who achieved a CR or PR
Time to Response (TTR) | Up to 30 months
  TTR is defined as the period of time from the date of first study drug administration until the first objective documentation of a CR or PR per RECIST 1.1.
Time to Progression (TTP) | Up to 30 months
  TTP is defined as the time from the date of first study drug administration until the start of disease progression per RECIST Version 1.1.
Progression Free Survival (PFS) | Up to 54 months
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression per RECIST 1.1. or death due to any cause
Overall Survival (OS) | Up to 54 months
  OS is defined as the time from first dose of study treatment to the date of death, irrespective of the cause of death
PK parameter: Area under the plasma concentration time curve (AUC) | Cycle 1 (28 days)
  Characterization of the PK profile of FHD-286
Plasma concentration vs. time profiles | Cycle 1 (28 days)
  Plasma concentration of FHD-286 at the scheduled timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Reilly, MD, Study Director — Foghorn Therapeutics
Locations (11):
- United States (9):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Miami Health System, Sylvester Comprehensive Cancer Center, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sidney Kimmel Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Institute Curie Hospital, Paris, France
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No